CLINICAL TRIAL: NCT04242537
Title: A Randomized Control Trial to Assess the Effectiveness of Apneic Oxygenation in Adults Using Low Flow or High Flow Nasal Cannula With Head Side Elevation Compared With Usual Care to Prevent Desaturation During Endotracheal Intubation
Brief Title: Apneic Oxygenation in the Emergency Department
Acronym: ApOxED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Shahan Waheed, Principal investigator and Consultant Emergency Medicine, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 192002ER-PK
Record Dates: First submitted 2020-01-19; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Apneic Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High flow oxygen delivery (Experimental): Oxygen delivery with high flow nasal cannula with head side elevation to 30 degrees
  Interventions: Device: High flow nasal cannula oxygen delivery
- Low Flow oxygen delivery (Experimental): Low flow oxygen delivery through nasal cannula with head side elevation to 30 degrees
  Interventions: Device: Low flow nasal cannula oxygen delivery
- Standard practice of care (No Intervention): No oxygen delivery either high flow or low flow through nasal cannula

INTERVENTIONS:
Device: High flow nasal cannula oxygen delivery — It includes the delivery of oxygen through a high flow nasal cannula with head side elevation to 30 degrees to prevent desaturation and improve first pass success rate of endotracheal intubation
  Other Names: High Flow nasal cannula
  Arms: High flow oxygen delivery
Device: Low flow nasal cannula oxygen delivery — It includes the delivery of oxygen through a low flow nasal cannula coupled with head side elevation to 30 degrees to prevent desaturation and improve first pass success rate of endotracheal intubation
  Other Names: Low Flow nasal cannula
  Arms: Low Flow oxygen delivery

SUMMARY:
Apneic oxygenation is a process of delivering continuous oxygen during direct laryngoscopy. Nasal cannulas are used for the purpose of oxygenation; for delivering either low flow or high flow oxygen but haven't been tested in terms of a superior study design on improving patient outcomes. In this study the investigators propose to assess the effect of giving low flow oxygen with head side elevation versus high flow oxygen with head side elevation against the usual practice of care in which no oxygen is provided during direct laryngoscopy on participant's oxygenation level. This will be a three arm study instituting block randomization technique. There will be no blinding due to the nature of intervention. The primary outcomes are lowest non-invasive oxygen saturation measurement during direct laryngoscopy and two minutes after the placement of the tube and first pass success rate. The intervention is unique as the investigators have introduced head side elevation up to 30 degrees for improving glottis visualization and low or high flow oxygen delivery on grounds to improve oxygenation for patient safety undergoing endotracheal intubation. The technique if proved successful can be employed as a method of airway management in the emergency room. The results of the study will open new horizons for the development of guidelines to utilize it as a routine measure, during airway management in the emergency room.

DETAILED DESCRIPTION:
Intervention (High Flow and Low Flow):

The participants after fulfilling the eligibility criteria will be randomly assigned to the respective arm (High Flow, Low Flow or Standard). For procedure, depending upon the arm, the head side of the patient bed will be elevated up to 30 degrees in order to better visualize the glottis. The participants in the high flow oxygen delivery through nasal cannula preoxygenation will be set for 4 min at 6 L/min through humidified and heated pure oxygen (fraction of inspired oxygen 100%, 37C). Similarly, participant in the low flow oxygen delivery through nasal cannula preoxygenation will be set for 4 min at 3 L/min through humidified and heated pure oxygen (faction of inspired oxygen 100%, 37C). Throughout the procedure the high flow nasal cannula or low flow nasal cannula will be maintained trying to achieve a continuous oxygen during direct laryngoscopy for RSI.

Standard Arm:

In the standard arm the head end of the bed will not be raised to 30 degrees instead the whole bed is raised up to the operator belly button in order to ease glottis visualization. In the standard group the preoxygenation is for 4 min or till achievement of peripheral oxygen saturation greater than 95% with a face mask that will be connected to the oxygen port at 10 L/min. During the direct laryngoscopy there will be no insufflation of oxygen through nasal cannula or face mask.

Data collection:

Research staff involved in collecting data, will be independent from primary research team in order to minimize observer bias. The oxygen saturations will be recorded using pulse oximetry (through a standard infrared oximetry tape) exclusively used for research purpose and will record time using stop watch (Casio Digital Stop Watch) during and after the procedure. The operator will report research staff about all subjective assessments of difficult intubation and airway complications during procedure on the data collection tool. The operator while performing the direct laryngoscopy, if experience difficulty as per Corkman Lehman grade, will inform research staff for protocol deviation.

Intubation attempts (number of time laryngoscope blade placed in the mouth) will be counted for each patient. In those patients where first pass is failed and subsequent attempt is made without assisted ventilation, the apnea time will be noted as mentioned above. To confirm the accuracy of data collected, the investigators will conduct a concurrent assessment of the outcomes for a convenience sample of 10% of enrolled participants.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18 years and above) requiring endotracheal intubation in the emergency department.
2. Intubation performed by the emergency medicine physician who are post graduate trainee year IV and above. The year IV and above cut off is taken because at this time the trainees have done more than 20 endotracheal intubations. The operators are assessed through direct supervision and confirmation through filing of their procedural log books

Exclusion Criteria:

1. Supervisor or operator feels specific intra-procedural oxygenation technique will be required.
2. Patients presenting with cardiac arrest
3. Pregnant patients (as the patients are at risk of aspiration and high oxygen delivery can have bad outcomes on the fetus)
4. Patients with 'Do not resuscitate' order.
5. Morbidly obese on assessment as such patient may need pre intubation preparation of the head side and more controlled settings.
6. Patient who are shifted from another hospital post intubation
7. Patients with interstitial lung disease or lung tumor
8. Neck trauma (expanding neck hematoma)
9. Neck and Oral cavity cancers, or patients with cancers of the neck and oral cavity who have undergone surgery, post radiation of the neck and oral cavity cancers.
10. Pulse oximetry <90% in ambient air.
11. Body mass index > 35kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Lowest noninvasive oxygenation value | Within 3 hours, beginning from the administration of the sedation or the neuromuscular blocker till the placement of the endotracheal tube
  The lowest noninvasive oxygenation value in any time between administration of sedation and/or neuromuscular blockade to successful endotracheal intubation
First pass success rate | With in 3 hours of the start of procedure for placement of endotracheal tube
  Single successful attempt for the placement of endotracheal tube in the trachea during direct laryngoscopy and subsequent confirmation.

SECONDARY OUTCOMES:
Safe Apnea Time | With in 3 hours beginning from the administration of the sedation and or neuromuscular blockade drug to the placement of the endotracheal tube
  the time from the administration of sedation and/or neuromuscular blockade to success to successful endotracheal intubation (safe apnea time)
Direct laryngoscopy grades | During the endotracheal tube placement
  Grade of largyogoscopic view as per Corkman Lehane Laryngoscopic grades (Grade I to IV) on first attempt.
Nonhypoxia complications | 6 hours starting from the endotracheal tube placement.
  Incidence of non-hypoxia complications (e.g. arrhythmia, hypotension, tracheal rupture, vocal cord injury)
Tube malposition | 6 hours starting from the endotracheal tube placement.
  Incidence of post-intubation tube malposition on Chest X ray

REFERENCES:
- [Derived] Waheed S, Kapadia NN, Jawed DR, Raheem A, Khan MF. Randomized controlled trial to assess the effectiveness of apnoeic oxygenation in adults using a low-flow or high-flow nasal cannula with head side elevation during endotracheal intubation in the emergency department. BMC Res Notes. 2025 Jul 1;18(1):264. doi: 10.1186/s13104-025-07328-7. PMID 40598378
- [Derived] Waheed S, Kapadia NN, Khan MF, Kerai SM, Raheem A, Naeem R. Randomised controlled trial to assess the effectiveness of apnoeic oxygenation in adults using low-flow or high-flow nasal cannula with head side elevation versus usual care to prevent desaturation during endotracheal intubation in the emergency department (ApOxED): study protocol. BMJ Open. 2020 Nov 16;10(11):e037964. doi: 10.1136/bmjopen-2020-037964. PMID 33199418